CLINICAL TRIAL: NCT00584129
Title: Determining the Efficacy of Pre-treatment Swallowing Therapy as a Means to Improve Dysphagia Quality of Life When Compared to Post-Treatment Therapy.
Brief Title: Pre-treatment Exercises Versus Post-treatment Exercises for Dysphagia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: American Academy of Otolaryngology-Head and Neck Surgery Foundation (Other)
Responsible Party: Principal Investigator, William Carroll, MD, Professor of Surgery, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: F060123002; F060123002
Record Dates: First submitted 2007-12-21; First posted 2008-01-02 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Head and Neck Cancer
Keywords: Cancer; Dysphagia; Radiation; Patients with H&N cancer who will be receiving chemoradiation
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms; Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Patients will receive pre-treatment swallowing exercises.
  Interventions: Other: Pre-treatment swallowing exercises
- 2 (Active Comparator): Post-treatment swallowing exercises.
  Interventions: Other: Post-treatment swallowing exercises.

INTERVENTIONS:
Other: Pre-treatment swallowing exercises — Swallowing exercises will be started pre-treatment with radiation.
  Arms: 1
Other: Post-treatment swallowing exercises. — Patients to start swallowing exercises after completion of radiation therapy.
  Arms: 2

SUMMARY:
The purpose of this project is to determine if pre-treatment swallowing exercises can improve post-treatment swallowing function in patients undergoing radiation with or without chemotherapy for advanced squamous cell carcinoma of the head and neck.

ELIGIBILITY:
Inclusion Criteria:

* Stage III or IV squamous cell cancer of teh pharynx and larynx
* Patients who will be receiving chemoradiation
* Age 19 years of age or older
* Must sign informed consent.

Exclusion Criteria:

* Prior cancer diagnosis
* Metastatic disease
* Cognitive Impairment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2006-02; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
To test whether pre-treatment swallowing exercises compared with "usual care" (where exercises are taught post-treatment) improves quality of life in patients undergoing chemoradiation therapy for advanced head and neck cancer. | 8 weeks, 6 months, 12 months post radiation treatment

SECONDARY OUTCOMES:
To test whether pre-treatment swallowing exercises compared with usual care improves secondary outcome measures related to dysphagia in this patient population. | 8 weeks, 6 mnths and 12 months post radiation.

CONTACTS AND LOCATIONS:
Overall Officials: William R. Carroll, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Division of Otolaryngology, Birmingham, Alabama, United States